CLINICAL TRIAL: NCT07319910
Title: Tumor Treating Fields (TTFields, 150kHz) Concomitant With Gemcitabine and Nab-paclitaxel for Front-line Treatment of Locally Advanced Pancreatic Adenocarcinoma: EF-54/PANOVA-3CA
Brief Title: Continued Access Program for Tumor Treating Fields (TTFields) Used With Chemotherapy (Gemcitabine and Nab-Paclitaxel) in Adults With Locally Advanced Pancreatic Cancer (PANOVA-3CA)
Acronym: PANOVA-3CA
Status: Temporarily not available | Type: Expanded Access
Sponsor: NovoCure GmbH (Industry)
Responsible Party: Sponsor
Organization: NovoCure Ltd. (Industry)
Other Study IDs: EF-54
Record Dates: First submitted 2025-12-18; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; Taxes

INTERVENTIONS:
Device: TTFields — TTFields is a non-invasive locoregional therapy that uses alternating electric fields. TTFields are delivered to the abdomen though adhesive transducer arrays connected to the NovoTTF-200T system.
Drug: Gemcitabine — per standard of care
Drug: Nab paclitaxel — per standard of care

SUMMARY:
The EF-54 program (PANOVA-3CA) is a continued access program for adults with locally advanced pancreatic cancer to access TTFields therapy in combination with gemcitabine and nab-paclitaxel. The purpose of the program is to allow eligible patients to have access to TTFields while the NovoTTF-200T system is under FDA review. Safety and device performance will be monitored during routine clinical care.

DETAILED DESCRIPTION:
This is a non-comparative continued access program. All enrolled patients who meet eligibility criteria will receive TTFields with gemcitabine and nab-paclitaxel.

Eligible patients are ≥22 years old, have histologically or cytologically confirmed de novo pancreatic adenocarcinoma not amenable to surgical resection and without evidence of distant metastases, an ECOG performance status of 0-2, and are candidates for gemcitabine plus nab-paclitaxel chemotherapy.

Patients will continue TTFields therapy in combination with chemotherapy according to the treating physician's and site's local standard of care until local disease progression is identified. After discontinuation, subsequent care and follow-up are per treating physician's and site's local standard. There is no protocol defined post-treatment assessments mandated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 22 years
* Histologically or cytologically confirmed de novo pancreatic adenocarcinoma
* Locally advanced, non-metastatic disease
* ECOG performance status of 0-2
* Candidate for treatment with gemcitabine and nab-paclitaxel
* Able to operate the NovoTTF-200T system independently or with caregiver support

Exclusion Criteria:

* Prior palliative treatment to the pancreatic tumor
* Other active malignancies within the past 5 years (except certain early-stage cancers)
* Significant uncontrolled medical conditions or infections that would interfere with therapy
* Implantable electronic devices in the torso
* Known severe hypersensitivity to adhesives, hydrogel, or chemotherapy agents
* Pregnancy or breastfeeding

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult